CLINICAL TRIAL: NCT06358079
Title: Isolated Cardiotomy Circuit for Re-infusion of Unwashed Shed Blood During Off-pump Coronary Artery Surgery
Brief Title: Re-infusion of Unwashed Shed Blood During Off-pump Surgery
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Damascus University (Other)
Responsible Party: Principal Investigator, Mohammad Bashar Izzat, Professor, Damascus University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 258
Record Dates: First submitted 2024-03-27; First posted 2024-04-10 (Actual); Last update posted 2024-04-10 (Actual); Status verified 2024-04

CONDITIONS: Coronary Artery Disease; Blood Transfusion Complication; Cardiovascular Complication
Keywords: surgery; coronary artery bypass grafting; blood; off-pump; auto-transfusion
MeSH Terms: conditions — Coronary Artery Disease; Transfusion Reaction

STUDY DESIGN:
Intervention Model Description: A prospective study involving patients undergoing off-pump coronary artery bypass surgery. Patients will be randomized to two groups; an isolated cardiotomy circuit for re-infusion of unwashed shed blood will be used in group (a) and the conventional no re-infusion technique will be used in group (b).
Who Masked: Outcomes Assessor
Masking Description: Outcome assessor will be blinded to the group type when analyzing data
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group 1: Use of circuit (Experimental): Re-infusion of unwashed shed blood
  Interventions: Procedure: Re-infusion of unwashed shed blood
- Group 2: No circuit (No Intervention): No re-infusion of unwashed shed blood

INTERVENTIONS:
Procedure: Re-infusion of unwashed shed blood — Use of an isolated cardiotomy circuit for re-infusion of unwashed shed blood during off-pump coronary artery surgery
  Arms: Group 1: Use of circuit

SUMMARY:
To assess the efficacy and side-effects of re-infusion of unwashed shed blood during off-pump coronary artery surgery using a novel cardiotomy circuit.

DETAILED DESCRIPTION:
Introduction Blood transfusion is often required during cardiac surgical operations, and may be associated with known risks and complications. Off-pump coronary artery surgery has been shown to be associated with reduced need for blood transfusion, and cell-savers are widely used as an additional method for reducing blood transfusion demands.

Auto-transfusion of unwashed suctioned blood intra-operatively is thought to increase the inflammatory response and infective complications, but data related to this approach are scares.

Aims

To assess the effects and benefits of using an isolated cardiotomy circuit for re-infusion of unwashed shed blood during off-pump surgery and compare it to the conventional no re-infusion technique. Assessments will focus on:

* clinical outcome
* transfusion requirements
* inflammatory response
* alveolar/arterial oxygen pressure gradients
* cognitive status
* cost-benefit

Study design A prospective study involving patients undergoing off-pump coronary artery bypass surgery. Patients will be randomized to two groups; an isolated cardiotomy circuit for re-infusion of unwashed shed blood will be used in group (a) and the conventional no re-infusion technique will be used in group (b).

Participants Patients undergoing off-pump coronary artery bypass surgery.

Setting Damascus University Cardiac Surgery Hospital

ELIGIBILITY:
Inclusion Criteria:

* All patients undergoing isolated off-pump coronary artery bypass surgery between March 1st, 2024 and March 31st, 2026.

Exclusion Criteria:

* Missing data.
* Patients outside the study period.
* Patients under the age of 40 years or over the age of 75 years.
* Patients with impaired left ventricular function (EF less the 40%).
* Patients with history of renal failure, hepatic failure, CVA, or TIA.
* Patients who have not stopped anticoagulants (except aspirin) for 4 days preoperatively.
* Emergency operations.

Ages: 40 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2024-03-27 (Actual); Primary Completion 2026-03-30 (Estimated); Study Completion 2026-03-30 (Estimated)

PRIMARY OUTCOMES:
blood transfusion requirements | up to 5 days post-operatively
  volume of blood (ml) transfused
inflammatory response | pre-operatively, immediately post-operatively, and 24 hours post-operatively
  changes in IL-6
alveolar/arterial oxygen pressure gradients | pre-, 4 hours post-operatively, and post-extubation
  changes in alveolar/arterial oxygen pressure gradients peri-operatively
cost-benefit | up to 5 days postoperatively
  cost of blood products, circuits and hospital stay
Neuro-markers | pre-operatively, immediately post-operatively, and 24 hours post-operatively
  Changes in S-100
myocardial marker CK-MB | pre-operatively, immediately post-operatively, and 24 hours post-operatively
  changes in CK-MB
myocardial marker troponin-I | pre-operatively, immediately post-operatively, and 24 hours post-operatively
  changes in troponin-I
blood loss | up to 24 hours post-operatively
  volume (ml) of blood lost
complement response | pre-operatively, immediately post-operatively, and 24 hours post-operatively
  changes in C3a

CONTACTS AND LOCATIONS:
Overall Officials: Mohammad Bashar Izzat, FRCS(CTh), Study Chair — Damascus University
Locations (1):
- Damascus University Cardiac Surgery Hospital, Damascus, Syria

IPD SHARING:
Plan to Share IPD: Yes
Data will be deposited in a Data Repository
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: Upon completion of the study and will be there permanently
Access Criteria: Open to all

REFERENCES:
- [Background] Liumbruno GM, Waters JH. Unwashed shed blood: should we transfuse it? Blood Transfus. 2011 Jul;9(3):241-5. doi: 10.2450/2011.0109-10. Epub 2011 Apr 20. No abstract available. PMID 21627923
- [Background] Konig G, Waters JH. Washing and filtering of cell-salvaged blood - does it make autotransfusion safer? Transfus Altern Transfus Med. 2012 Dec 1;12(3-4):78-87. doi: 10.1111/j.1778-428X.2012.01155.x. No abstract available. PMID 24955005
- [Background] Westerberg M, Gabel J, Bengtsson A, Sellgren J, Eidem O, Jeppsson A. Hemodynamic effects of cardiotomy suction blood. J Thorac Cardiovasc Surg. 2006 Jun;131(6):1352-7. doi: 10.1016/j.jtcvs.2005.12.067. PMID 16733169
- [Background] Gabel J, Westerberg M, Bengtsson A, Jeppsson A. Cell salvage of cardiotomy suction blood improves the balance between pro- and anti-inflammatory cytokines after cardiac surgery. Eur J Cardiothorac Surg. 2013 Sep;44(3):506-11. doi: 10.1093/ejcts/ezt019. Epub 2013 Feb 12. PMID 23404689
- [Background] Yasukawa T, Manabe S, Hiraoka D, Hirayama D, Kinoshita R, Komori M, Hosokawa M, Hirooka K. Safety and efficacy of a simple cardiotomy suction system as a blood salvage procedure during off-pump coronary artery bypass surgery. J Artif Organs. 2019 Sep;22(3):194-199. doi: 10.1007/s10047-019-01103-9. Epub 2019 Apr 9. PMID 30968273
- [Background] Vu T, Smith JA. An Update on Postoperative Cognitive Dysfunction Following Cardiac Surgery. Front Psychiatry. 2022 Jun 15;13:884907. doi: 10.3389/fpsyt.2022.884907. eCollection 2022. PMID 35782418
- [Background] Dabrowski W, Rzecki Z, Czajkowski M, Pilat J, Wacinski P, Kotlinska E, Sztanke M, Sztanke K, Stazka K, Pasternak K. Volatile anesthetics reduce biochemical markers of brain injury and brain magnesium disorders in patients undergoing coronary artery bypass graft surgery. J Cardiothorac Vasc Anesth. 2012 Jun;26(3):395-402. doi: 10.1053/j.jvca.2011.10.014. Epub 2011 Dec 28. PMID 22206712
- [Background] Allen SJ, McBride WT, McMurray TJ, Phillips AS, Penugonda SP, Campalani G, Young IS, Armstrong MA. Cell salvage alters the systemic inflammatory response after off-pump coronary artery bypass grafting surgery. Ann Thorac Surg. 2007 Feb;83(2):578-85. doi: 10.1016/j.athoracsur.2006.09.041. PMID 17257991
- [Background] Baker RA, Merry AF. Cell salvage is beneficial for all cardiac surgical patients: arguments for and against. J Extra Corpor Technol. 2012 Mar;44(1):P38-41. PMID 22730871
- [Background] Cote CL, Yip AM, MacLeod JB, O'Reilly B, Murray J, Ouzounian M, Brown CD, Forgie R, Pelletier MP, Hassan A. Efficacy of intraoperative cell salvage in decreasing perioperative blood transfusion rates in first-time cardiac surgery patients: a retrospective study. Can J Surg. 2016 Sep;59(5):330-6. doi: 10.1503/cjs.002216. PMID 27668331
- [Background] Engels GE, van Klarenbosch J, Gu YJ, van Oeveren W, de Vries AJ. Intraoperative cell salvage during cardiac surgery is associated with reduced postoperative lung injury. Interact Cardiovasc Thorac Surg. 2016 Mar;22(3):298-304. doi: 10.1093/icvts/ivv355. Epub 2015 Dec 23. PMID 26705299
- [Background] Izzat MB, Almohammad F, Raslan AF. Off-pump grafting does not reduce postoperative pulmonary dysfunction. Asian Cardiovasc Thorac Ann. 2017 Feb;25(2):113-117. doi: 10.1177/0218492316689350. Epub 2017 Jan 13. PMID 28084083
- [Background] Wan IY, Arifi AA, Wan S, Yip JH, Sihoe AD, Thung KH, Wong EM, Yim AP. Beating heart revascularization with or without cardiopulmonary bypass: evaluation of inflammatory response in a prospective randomized study. J Thorac Cardiovasc Surg. 2004 Jun;127(6):1624-31. doi: 10.1016/j.jtcvs.2003.10.043. PMID 15173716
- [Background] Kim KI, Lee WY, Ko HH, Kim HS, Jeong JH. Hemoglobin Level to Facilitate Off-Pump Coronary Artery Bypass without Transfusion. Korean J Thorac Cardiovasc Surg. 2014 Aug;47(4):350-7. doi: 10.5090/kjtcs.2014.47.4.350. Epub 2014 Aug 5. PMID 25207243
- [Background] Kitano T, Hattori S, Miyakawa H, Yoshitake S, Iwasaka H, Noguchi T. Unwashed shed blood infusion causes deterioration in right ventricular function after coronary artery surgery. Anaesth Intensive Care. 2000 Dec;28(6):642-5. doi: 10.1177/0310057X0002800605. PMID 11153289
- [Background] Munoz M, Slappendel R, Thomas D. Laboratory characteristics and clinical utility of post-operative cell salvage: washed or unwashed blood transfusion? Blood Transfus. 2011 Jul;9(3):248-61. doi: 10.2450/2010.0063-10. Epub 2010 Sep 14. No abstract available. PMID 21084005
- [Background] Murphy GJ, Rogers CS, Lansdowne WB, Channon I, Alwair H, Cohen A, Caputo M, Angelini GD. Safety, efficacy, and cost of intraoperative cell salvage and autotransfusion after off-pump coronary artery bypass surgery: a randomized trial. J Thorac Cardiovasc Surg. 2005 Jul;130(1):20-8. doi: 10.1016/j.jtcvs.2004.12.006. PMID 15999036
- [Background] Roman MA, Abbasciano RG, Pathak S, Oo S, Yusoff S, Wozniak M, Qureshi S, Lai FY, Kumar T, Richards T, Yao G, Estcourt L, Murphy GJ. Patient blood management interventions do not lead to important clinical benefits or cost-effectiveness for major surgery: a network meta-analysis. Br J Anaesth. 2021 Jan;126(1):149-156. doi: 10.1016/j.bja.2020.04.087. Epub 2020 Jun 30. PMID 32620259
- [Background] Wan S, Izzat MB, Lee TW, Wan IY, Tang NL, Yim AP. Avoiding cardiopulmonary bypass in multivessel CABG reduces cytokine response and myocardial injury. Ann Thorac Surg. 1999 Jul;68(1):52-6; discussion 56-7. doi: 10.1016/s0003-4975(99)00315-x. PMID 10421114
- [Background] Vieira SD, da Cunha Vieira Perini F, de Sousa LCB, Buffolo E, Chaccur P, Arrais M, Jatene FB. Autologous blood salvage in cardiac surgery: clinical evaluation, efficacy and levels of residual heparin. Hematol Transfus Cell Ther. 2021 Jan-Mar;43(1):1-8. doi: 10.1016/j.htct.2019.08.005. Epub 2019 Nov 7. PMID 31791879
- [Background] Wozniak MJ, Sullo N, Qureshi S, Dott W, Cardigan R, Wiltshire M, Morris T, Nath M, Bittar N, Bhudia SK, Kumar T, Goodall AH, Murphy GJ. Randomized trial of red cell washing for the prevention of transfusion-associated organ injury in cardiac surgery. Br J Anaesth. 2017 May 1;118(5):689-698. doi: 10.1093/bja/aex083. PMID 28475670